CLINICAL TRIAL: NCT07065955
Title: Effects of the Longevity Diet and the Fasting-mimicking Diet on Body Composition, Risk Factors for Age-related Diseases
Brief Title: Longevity Diet and the Fasting-mimicking Diet
Status: Completed | Type: Observational
Sponsor: Fondazione Valter Longo (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-UCALPRG-0082112
Record Dates: First submitted 2025-03-17; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Overweight; Obesity; Metabolic Syndrome; Autoimmune Diseases; Inflammatory Disease; Health, Subjective
Keywords: Longevity; Fasting Mimicking Diet; Longevity Diet; Diet; Aging; FMD; Nutrition; Diseases; Clinical Trial; Fat Mass; Phase Angle; Muscle Mass; Caloric Restriction
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Autoimmune Diseases; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Longevity diet alone or in combination with fasting mimicking diet — The longevity diet generally consists of three isocaloric meals and one snack (for normal-weight individuals) or slightly hypocaloric meals (in the case of overweight or obesity). The diet consists of 50-60% of calories from complex carbohydrates, 30-35% of calories from mostly unsaturated fats, and 10-11% of calories from proteins, primarily from plant sources and fish, and occasionally from eggs, dairy, and meat, especially for those over 65. The diet is formulated to provide all necessary nutrients, including vitamins and minerals. The fasting-mimicking diet is a dietary intervention in which normal food is replaced with a standardized, highly hypocaloric vegan diet for a limited period of 5 consecutive days. This diet is designed to stimulate the same processes normally activated during fasting while minimizing the side effects of total food deprivation.

SUMMARY:
This retrospective clinical study examines the impact of the longevity diet and fasting-mimicking diet (FMD), either alone or combined, on body composition and health indicators. Focused on subjects from the Valter Longo Foundation (2019-2024), the study aims to evaluate their effects on body fat percentage, lean mass, muscle function, and lipid profiles.

The longevity diet, rooted in centenarian dietary traditions, emphasizes isocaloric meals with a balance of complex carbohydrates, unsaturated fats, and plant-based proteins. FMD involves a 5-day highly hypocaloric vegan diet to simulate fasting benefits. Hypothesizing that a return to a modified Mediterranean diet or incorporating FMD could improve overall health, the study spans diverse cohorts based on intervention type, duration, obesity level, and physio-pathological status.

Data, collected from electronic medical records, will undergo statistical analyses to compare pre- and post-intervention measurements, exploring outcomes across subgroups. Ethical considerations, including de-identified data and informed consent, ensure compliance with clinical research regulations.

In conclusion, this study provides valuable insights into the potential health and longevity benefits of the longevity diet and FMD, with implications for public wellness.

DETAILED DESCRIPTION:
1. Introduction Aging is often accompanied by numerous chronic degenerative conditions that compromise the quality of life and lead to dependency. However, a favorable interaction between genetic and environmental factors could lead to a significantly higher life expectancy, free from conditions that significantly compromise both the quality and duration of life, highlighting that increased longevity is not necessarily accompanied by one or more pathological conditions.

   It is widely accepted that the quality and quantity of nutrition are essential factors in maintaining health and preventing diseases. Making healthy and conscious dietary choices can indeed alter the course of life in terms of both duration and health.

   Numerous epidemiological studies have demonstrated the critical role of a proper dietary regimen in the risk of developing age-related diseases. Furthermore, recent studies have highlighted how short periods of extreme calorie reduction with adequate nutrient intake (5 days, fasting-mimicking diet, FMD) can impact metabolism, producing numerous beneficial effects in both healthy individuals and those with chronic degenerative conditions such as cancer, cardiovascular diseases, diabetes, and autoimmune diseases.

   Theories about senescence usually focus on the aging process and not on the ability of organisms to stay young. The longevity diet proposed in this study is intended to be effective in achieving the goal of extending youth for as long as possible, optimizing protection, regeneration, and rejuvenation while minimizing diseases. It is based on five pillars that support the scientific evidence of the program: basic research, epidemiology, clinical studies, centenarian studies, and complex systems studies.

   Essentially, the longevity diet incorporates the dietary tradition of healthy centenarians, characterized by simplicity and products typical of their region of origin.

   This type of diet generally consists of three isocaloric meals and one snack (for normal-weight individuals) or slightly hypocaloric meals (in the case of overweight or obesity). The diet consists of 50-60% of calories from complex carbohydrates, 30-35% of calories from mostly unsaturated fats, and 10-11% of calories from proteins, primarily from plant sources and fish, and occasionally from eggs, dairy, and meat, especially for those over 65. The diet is formulated to provide all necessary nutrients, including vitamins and minerals.

   The fasting-mimicking diet is a dietary intervention in which normal food is replaced with a standardized, highly hypocaloric vegan diet for a limited period of 5 consecutive days. This diet is designed to stimulate the same processes normally activated during fasting while minimizing the side effects of total food deprivation.

   This retrospective clinical study aims to investigate the two different approaches: the longevity diet and the fasting-mimicking diet, to assess both their feasibility and effectiveness when used individually or in combination.

   1.1 Background and Hypotheses The Italian population has moved away from the traditional Mediterranean diet and now predominantly follows a Western-style diet that is hypercaloric, rich in saturated fats, animal protein, and sugars. We hypothesize that a return to the original Mediterranean diet with modifications based on the scientific evidence of recent decades (longevity diet), and/or short periods of fasting-mimicking diet (5 days), can improve the overall health conditions of the population.
2. Objectives and Purpose of the Study Primary Objective: To evaluate whether the longevity diet and the fasting-mimicking diet, either individually or in combination, can reduce the percentage of body fat in a cohort of subjects stratified by gender, age, body mass index, and defined physio-pathological states.

   Secondary Objectives: To assess whether the longevity diet and the fasting-mimicking diet, either individually or in combination, can positively influence parameters related to the general health status of the analyzed sample, including (i) percentage of lean mass, (ii) phase angle as an indirect indicator of muscle function and cellular integrity, (iii) waist and hip circumference, (iv) total cholesterol, HDL, and LDL.
3. Study Design This is a retrospective, observational, single-center study to evaluate the effect of specific nutritional interventions (fasting-mimicking diet (FMD) and longevity diet (LD)) on reducing body fat. To achieve this, retrospective data from bioimpedance, anthropometric, and clinical analyses of subjects who underwent at least one of the two nutritional interventions (individually or in combination) at the Valter Longo Foundation in Milan from 2019 to 2024 will be analyzed. In particular, information from subjects who underwent at least two nutritional visits with bioimpedance analysis with a gap of at least 3 months between them will be considered. The subjects will be characterized based on (i) the type of nutritional intervention (FMD only, LD only, or combinations of LD and FMD); (ii) the duration of the nutritional intervention (short, medium, or long); (iii) the degree of obesity (normal weight, overweight, and obese); and (iv) physio-pathological status.
4. Data Collection and Analysis Data will be collected retrospectively from the electronic medical records of the Valter Longo Foundation. Bioimpedance analysis, anthropometric measurements, and clinical parameters including lipid profiles will be used to assess changes in body composition, body fat percentage, lean mass percentage, phase angle, waist circumference, hip circumference, and blood lipid levels.
5. Statistical Analysis Statistical analyses will be performed using appropriate statistical software packages. Descriptive statistics will be used to summarize baseline characteristics, and paired t-tests or non-parametric equivalents will be used to compare pre- and post-intervention measurements. Analysis of variance will be used to compare outcomes across different subgroups based on type of intervention, duration, degree of obesity, and physio-pathological status. Correlation analyses may also be performed to explore associations between changes in body composition and other variables. A p-value of less than 0.05 will be considered statistically significant.
6. Ethical Considerations This study will be conducted in accordance with ethical principles and regulations governing clinical research. All data will be de-identified and handled in compliance with data protection regulations. Informed consent will be obtained from all subjects included in the study.
7. Conclusion This retrospective clinical study aims to investigate the effects of the longevity diet and the fasting-mimicking diet, either individually or in combination, on body composition, age-related disease risk factors, and aging markers. The study will provide valuable insights into the potential benefits of these dietary interventions in promoting health and longevity, which could have significant implications for public health and wellness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients and/or those with diseases, excluding neoplastic and neurodegenerative pathologies;
* Age >/= 18 years;
* Body mass index >/= 18.5 kg/m2;
* At least two visits, both characterized by bioimpedance and anthropometric analysis;
* At least 3 months between the first and last bioimpedance and anthropometric analysis;
* Signature of informed consent and privacy for the conducted visits.

Exclusion Criteria:

* Age < 18 years;
* Lack of informed consent or privacy;
* Women who are pregnant or breastfeeding;
* Patients affected by oncological and/or neurodegenerative pathologies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The bioimpedance, anthropometric, and clinical data of subjects who underwent at least one of the two nutritional interventions (individually or in combination) at the Valter Longo Foundation in Milan from 2019 to 2024 will be retrospectively analyzed. As this is a purely observational (retrospective) study with purely descriptive objectives, a formal power analysis estimation has not been conducted. However, considering that the Valter Longo Foundation in Milan is a regional reference point, it is estimated that approximately 250 subjects will be recruited retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Fat mass in % | Comparison of Fat mass in % at baseline and after a period between 3 months (minimum) and 2 years (maximum)
  The percentage of the Fat Mass in measured through a Bioimpedance Analysis (BIA) or a caliper

SECONDARY OUTCOMES:
Phase Angle | Comparison of Phase Angle at baseline and after a period between 3 months (minimum) and 2 years (maximum)
  The Phase Angle in measured through a Bioimpedance Analysis (BIA) in degrees
Free Fat Mass in percent | Comparison of Free Fat Mass in percent at baseline and after a period between 3 months (minimum) and 2 years (maximum)
  The percentage of the Free Fat Mass in measured through a Bioimpedance Analysis (BIA) or caliper
Waist Circumference | Comparison of Waist Circumference at baseline and after a period between 3 months (minimum) and 2 years (maximum)
  The Waist circumference is measured through a anthropometric tape in cm
Hips Circumference | Comparison of Hips Circumference at baseline and after a period between 3 months (minimum) and 2 years (maximum)
  The Hips circumference is measured through a anthropometric tape in cm
Total Cholesterol | Comparison of Total Cholesterol maximum 6 months before the first consultation and maximum 6 months after the last consultation
  The Total Cholesterol is measured through blood samples analyzed in a private and sepatate laboratory (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Valter Longo Onlus, Milan, Italy

REFERENCES:
- [Background] Ley SH, Ardisson Korat AV, Sun Q, Tobias DK, Zhang C, Qi L, Willett WC, Manson JE, Hu FB. Contribution of the Nurses' Health Studies to Uncovering Risk Factors for Type 2 Diabetes: Diet, Lifestyle, Biomarkers, and Genetics. Am J Public Health. 2016 Sep;106(9):1624-30. doi: 10.2105/AJPH.2016.303314. Epub 2016 Jul 26. PMID 27459454
- [Background] Mahabir S, Willett WC, Friedenreich CM, Lai GY, Boushey CJ, Matthews CE, Sinha R, Colditz GA, Rothwell JA, Reedy J, Patel AV, Leitzmann MF, Fraser GE, Ross S, Hursting SD, Abnet CC, Kushi LH, Taylor PR, Prentice RL. Research Strategies for Nutritional and Physical Activity Epidemiology and Cancer Prevention. Cancer Epidemiol Biomarkers Prev. 2018 Mar;27(3):233-244. doi: 10.1158/1055-9965.EPI-17-0509. Epub 2017 Dec 18. PMID 29254934
- [Background] Yu E, Rimm E, Qi L, Rexrode K, Albert CM, Sun Q, Willett WC, Hu FB, Manson JE. Diet, Lifestyle, Biomarkers, Genetic Factors, and Risk of Cardiovascular Disease in the Nurses' Health Studies. Am J Public Health. 2016 Sep;106(9):1616-23. doi: 10.2105/AJPH.2016.303316. Epub 2016 Jul 26. PMID 27459449
- [Background] Li Y, Pan A, Wang DD, Liu X, Dhana K, Franco OH, Kaptoge S, Di Angelantonio E, Stampfer M, Willett WC, Hu FB. Impact of Healthy Lifestyle Factors on Life Expectancies in the US Population. Circulation. 2018 Jul 24;138(4):345-355. doi: 10.1161/CIRCULATIONAHA.117.032047. PMID 29712712
- [Background] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779
- [Background] Crupi AN, Haase J, Brandhorst S, Longo VD. Periodic and Intermittent Fasting in Diabetes and Cardiovascular Disease. Curr Diab Rep. 2020 Dec 10;20(12):83. doi: 10.1007/s11892-020-01362-4. PMID 33301104
- [Background] Fanti M, Mishra A, Longo VD, Brandhorst S. Time-Restricted Eating, Intermittent Fasting, and Fasting-Mimicking Diets in Weight Loss. Curr Obes Rep. 2021 Jun;10(2):70-80. doi: 10.1007/s13679-021-00424-2. Epub 2021 Jan 29. PMID 33512641
- [Background] Gallus S, Odone A, Lugo A, Bosetti C, Colombo P, Zuccaro P, La Vecchia C. Overweight and obesity prevalence and determinants in Italy: an update to 2010. Eur J Nutr. 2013 Mar;52(2):677-85. doi: 10.1007/s00394-012-0372-y. Epub 2012 May 27. PMID 22645105
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Mishra A, Mirzaei H, Guidi N, Vinciguerra M, Mouton A, Linardic M, Rappa F, Barone R, Navarrete G, Wei M, Brandhorst S, Di Biase S, Morgan TE, Ram Kumar S, Conti PS, Pellegrini M, Bernier M, de Cabo R, Longo VD. Fasting-mimicking diet prevents high-fat diet effect on cardiometabolic risk and lifespan. Nat Metab. 2021 Oct;3(10):1342-1356. doi: 10.1038/s42255-021-00469-6. Epub 2021 Oct 14. PMID 34650272
- [Background] Brandhorst S, Choi IY, Wei M, Cheng CW, Sedrakyan S, Navarrete G, Dubeau L, Yap LP, Park R, Vinciguerra M, Di Biase S, Mirzaei H, Mirisola MG, Childress P, Ji L, Groshen S, Penna F, Odetti P, Perin L, Conti PS, Ikeno Y, Kennedy BK, Cohen P, Morgan TE, Dorff TB, Longo VD. A Periodic Diet that Mimics Fasting Promotes Multi-System Regeneration, Enhanced Cognitive Performance, and Healthspan. Cell Metab. 2015 Jul 7;22(1):86-99. doi: 10.1016/j.cmet.2015.05.012. Epub 2015 Jun 18. PMID 26094889

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT07065955/Prot_SAP_ICF_000.pdf